CLINICAL TRIAL: NCT07115355
Title: Removable Uterine Compression Sutures (RUCS): Evaluation of Efficacy and Safety in Postpartum Hemorrhage
Brief Title: Evaluating the Safety and Efficacy of RUCS in PPH
Acronym: RUCS-PPH
Status: Completed | Type: Observational
Sponsor: Havva Betül Bacak (Other Government)
Responsible Party: Sponsor-Investigator, Havva Betül Bacak, Specialist in Obstetrics and Gynecology, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: GopRucs
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RUCS Group: This group includes women aged 18-45 who experienced postpartum hemorrhage and were treated with Removable Uterine Compression Sutures (RUCS) at Gaziosmanpaşa Training and Research Hospital between January 2020 and November 2024. All patients had complete medical records and underwent retrospective data analysis.
  Interventions: Procedure: Removable Uterine Compression Suture (RUCS)

INTERVENTIONS:
Procedure: Removable Uterine Compression Suture (RUCS) — Removable Uterine Compression Suture (RUCS) is a uterus-preserving surgical technique used to control postpartum hemorrhage (PPH) when medical management fails. The suture is placed in a way that allows for its removal after hemostasis is achieved, potentially reducing the risk of complications such as intrauterine synechiae. In this study, RUCS was applied to 11 patients following delivery-related hemorrhage.

SUMMARY:
This retrospective observational study aims to evaluate the efficacy and safety of Removable Uterine Compression Sutures (RUCS) in the surgical management of postpartum hemorrhage (PPH). Eleven patients who developed PPH and underwent RUCS between January 2020 and November 2024 at Gaziosmanpaşa Training and Research Hospital were included. The primary outcomes assessed were hemorrhage control and procedure-related complications. Data were collected from patient records and analyzed descriptively.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) remains one of the leading causes of maternal morbidity and mortality worldwide. When medical management is insufficient, surgical interventions become necessary. Removable Uterine Compression Sutures (RUCS) have been developed as a uterus-sparing surgical technique that may offer effective hemostasis with a potentially lower risk of complications such as intrauterine synechiae, when compared to traditional permanent suture methods.

This single-center retrospective observational case series evaluated 11 patients who experienced PPH and were treated with RUCS at the Obstetrics and Gynecology Clinic of Gaziosmanpaşa Training and Research Hospital between January 2020 and November 2024. Patients were included if they had complete medical records and underwent RUCS after delivery. Cases involving other surgical techniques or missing data were excluded.

Clinical data were extracted from hospital archives and electronic medical systems. All data were anonymized prior to analysis. Descriptive statistics were used, including means and standard deviations for continuous variables and frequencies for categorical variables.

The study aimed to assess both the efficacy of RUCS in controlling bleeding and its safety by monitoring postoperative complications such as intrauterine synechiae and uterine necrosis. Initial findings indicate 100% success in hemostasis with no observed major complications, suggesting that RUCS may be a safe and effective option in selected cases of postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 to 45 years Diagnosed with postpartum hemorrhage (PPH) following delivery Treated with Removable Uterine Compression Suture (RUCS) Delivery and treatment performed at Gaziosmanpaşa Training and Research Hospital RUCS performed between January 2020 and November 2024 Complete and accessible medical records

Exclusion Criteria:

Incomplete or missing medical records Use of alternative surgical techniques other than RUCS Patients outside the age range of 18-45 Cases not treated at Gaziosmanpaşa Training and Research Hospital Postpartum hemorrhage not managed with RUCS

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of women aged 18-45 who developed postpartum hemorrhage following delivery and were treated with Removable Uterine Compression Sutures (RUCS) at Gaziosmanpaşa Training and Research Hospital between January 2020 and November 2024. Only patients with complete and accessible medical records were included in this retrospective case series.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Hemostasis success rate following RUCS application | Within the first 24 hours post-procedure
  Successful control of postpartum bleeding without the need for additional surgical intervention, blood transfusion exceeding 4 units, or hysterectomy.

CONTACTS AND LOCATIONS:
Overall Officials: fatih irice, md, Study Chair — University of Health Sciences, Gaziosmanpaşa Training and Research Hospital
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No